CLINICAL TRIAL: NCT02234687
Title: A mGlu2/3 Agonist in the Treatment of PTSD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The original PI, Alexander Neumeister, left NYULMC. No data was analyzed.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-00609
Record Dates: First submitted 2014-09-03; First posted 2014-09-09 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Post-traumatic Stress Disorder
Keywords: post-traumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — pomaglumetad methionil; LY 2140023

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo, one dose
  Interventions: Drug: Placebo
- Pomaglumetad Methionil 40mg (Experimental): Pomaglumetad Methionil 40mg, one dose, one time
  Interventions: Drug: Pomaglumetad Methionil 40mg
- Pomaglumetad Methionil 160mg (Experimental): Pomaglumetad Methionil 160mg, one dose, one time
  Interventions: Drug: Pomaglumetad Methionil 160mg

INTERVENTIONS:
Drug: Pomaglumetad Methionil 160mg — Pomaglumetad Methionil 160mg, one dose, one time
  Other Names: LY2140023
  Arms: Pomaglumetad Methionil 160mg
Drug: Pomaglumetad Methionil 40mg — Pomaglumetad Methionil 40mg, one dose, one time
  Other Names: LY2140023
  Arms: Pomaglumetad Methionil 40mg
Drug: Placebo — Placebo, one dose, one time
  Arms: Placebo

SUMMARY:
In this study, we propose to employ a randomized, double-blind, placebo-controlled, outpatient clinical trial to test the efficacy, safety, and tolerability of a 160 mg and 40 mg challenge of the mGlu2/3 agonist pomaglumetad methionil relative to placebo in modulating fear-potentiated startle response and behavior in adults with post-traumatic stress disorder (PTSD) (N=30). Each participant will receive a single dose of the study drug (40 mg vs 160 mg vs placebo in a 1:1:1 ratio).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 60 years of age, any race
* Primary, current Axis I diagnosis of post traumatic stress disorder (PTSD) according to Diagnostic and Statistical Manual of Mental Disorders - IV (DSM-IV) criteria
* Able to provide written informed consent

Exclusion Criteria:

* Past or current presence of psychotic symptoms, or diagnosis of a lifetime psychotic disorder including schizophrenia, schizoaffective disorder, bipolar disorder
* History of moderate or severe traumatic brain injury (TBI) with loss of consciousness
* Lifetime history of seizure disorder
* Current diagnosis of obsessive-compulsive disorder (OCD)
* Current diagnosis of bulimia nervosa or anorexia nervosa; or substance use disorder
* Alcohol or drug abuse in the past 90 days, or dependence in the past year.
* Individuals with a cumulative lifetime history of intravenous substance abuse longer than 1 year.
* Severe dissociation, defined as a Clinician Administered Dissociative States Scale (CADSS) score greater than 60 at baseline
* Patients with creatinine clearance <60 milliliters (mL)/min (moderate renal impairment)
* Current pregnancy or breast feeding; medical conditions that could interfere with correct interpretation of study data, i.e., individuals with the following medical conditions will be excluded: cancer in the past year, stroke, heart attack, angina, neurological disease (multiple sclerosis, epilepsy, Parkinson's disease), central nervous system (CNS) lesions including TBI with loss of consciousness, dementing illness, and/or liver or kidney disease. Patients with QT interval >450 msec (males) and >470 msec (females).
* Participants who have started new medication regimen for PTSD within 3 months prior to study start and subjects taking fluoxetine
* Current suicidality defined by emergent Columbia Suicide Severity Rating Scale (CSSRS)-defined suicidal behavior, a suicidal ideation score of 5 (indicating active suicidal ideation with specific plan and some level of intent) or 4 (indicating active suicidal ideation with some intent to act, without specific plan) on the CSSRS or in the absence of a CSSRS suicidal ideation score of 5 or 4 or CSSRS-defined suicidal behavior, if the investigator determines the patient to have a significant short-term risk for a suicide attempt.
* Individuals with active suicidal risk, active self-mutilation or aggressive behavior with threatening behavior toward others within the past year, as judged by the Principal Investigator
* Pregnant or lactating women
* Legal and Financial: Current legal proceedings resulting from the traumatic events. People whose continued receipt of financial benefits is contingent upon maintaining PTSD symptoms or who are waiting for a decision concerning the receipt of financial benefits based upon PTSD symptoms

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-02-11 (Actual); Study Completion 2016-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Marmar, MD, Principal Investigator — NYU School of Medicine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No Outcome Measures Analyzed; Study Terminated
Pre-assignment Details: No Outcome Measures Analyzed; Study Terminated
Groups:
- 40 mg Poma; Placebo; 160 mg Poma: Study Terminated. No outcome measures were analyzed
Period: Overall Study
Arm/Group | 40 mg Poma | Placebo | 160 mg Poma
Started | 6 (Study Terminated. No outcome measures were analyzed) | 4 | 4
Completed | 0 (Study Terminated. No outcome measures were analyzed) | 0 | 0
Not Completed | 6 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 40 mg Poma | 160 mg Poma | Total
Number analyzed (Participants) | 6 | 4 | 4 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 4 | 14
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 7
  Male | 3 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Effect of 160mg and 40mg of Pomaglumetad Methionil
Description: To evaluate the effect of 160mg and 40mg challenge of the mGlu2/3 receptor agonist pomaglumetad methionil relative to placebo in mitigating fear-potentiated startle using the neutral-predictable-unpredictable fear-potentiated startle paradigm in adults with post-traumatic stress disorder (PTSD). The primary index of unpredictable fear will be the difference score between startle magnitude in safe and unpredictable conditions in the absence of the cue.
Time Frame: 6 months
Population: 10 patients were enrolled and data for these 10 patients was not analyzed. Assuming a 2-tailed test,power=0.80, alpha=0.05, a total sample size of 30 (10 per group) is required to detect a moderate differential effect size change of a 160mg or 40 mg dose of pomaglumated methionil relative to placebo.
Groups:
- Pomaglumetad Methionil 160mg: Pomaglumetad Methionil 160mg, one dose, one time Pomaglumetad Methionil 160mg: Pomaglumetad Methionil 160mg, one dose, one time
- Pomaglumetad Methionil 40mg: Pomaglumetad Methionil 40mg, one dose, one time Pomaglumetad Methionil 40mg: Pomaglumetad Methionil 40mg, one dose, one time
Arm/Group | Placebo | Pomaglumetad Methionil 160mg | Pomaglumetad Methionil 40mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Groups:
- Placebo: Placebo, one dose Placebo: Placebo, one dose, one time
Arm/Group | Placebo | Pomaglumetad Methionil 160mg | Pomaglumetad Methionil 40mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/6 | 0/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Pomaglumetad Methionil 160mg (N=4) | Pomaglumetad Methionil 40mg (N=4)
Vomiting after receiving medication (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
PTSD symptoms became worse after the study (General disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
10 patients were enrolled and data for these 10 patients was not analyzed because enrollment must reach a certain threshold for reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes